CLINICAL TRIAL: NCT05455060
Title: Evaluation of Clinical Efficacy and Pharmacological Mechanism of a Mixed Chinese Herbal Formula in Atopic Dermatitis Patients by Integrating Metabolomics and Pharmacokinetic Analysis
Brief Title: Effects of a Mixed Chinese Herbal Formula on Atopic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Yang Ming Chiao Tung University (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taipei Medical University (Other)
Responsible Party: Principal Investigator, YANG SIEN-HUNG, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202200262A3C602
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Chinese herbal formula; Clinical trial; Microbiota; Metabolomics analysis; Pharmacokinetic study
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese herbal formula (CHF) (Experimental): The patients in CHF group will take CHF capsules, 12 capsules (6 gm) twice a day, total 12 gm a day for 12 weeks, and the dosage will be modified according to patients' body weight. (3gm BID for 20kg≦BW<40kg; 1.5gm BID for BW<20kg)
  Interventions: Drug: Chinese herbal formula (CHF)
- Control (Placebo Comparator): The patients in control group will take the placebo capsules, which has the similar look, smell, and taste. The dosage, frequency, and duration are the same as CHF group, in which 12 capsules (6 gm) twice a day, total 12 gm a day for 12 weeks, and the dosage will be modified according to patients' body weight. (3gm BID for 20kg≦BW<40kg; 1.5gm BID for BW<20kg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chinese herbal formula (CHF) — Each CHF capsule, weighing 500mg, is composed of Xiao-Feng-San 200mg, Zhen-Ren-Huo-Ming-Yin 200mg, Dictamnus dasycarpus 50mg and Houttuynia cordata 50mg. Patients will take the medicine 2 times a day (6gm BID for BW≥40kg), for 12 weeks, and the dosage will be modified according to patients' body weight. (3gm BID for 20kg≦BW<40kg; 1.5gm BID for BW<20kg)
  Arms: Chinese herbal formula (CHF)
Drug: Placebo — The patients in control group will take the placebo capsules, which has the similar look, smell, and taste. The dosage, frequency, and duration are the same as CHF group.
  Arms: Control

SUMMARY:
The aim of this study is to investigate the clinical therapeutic effects of a mixed Chinese herbal formula (CHF) in treating atopic dermatitis (AD) based on its effects on cytokine levels and immune cell counts. Th1/Th2/Th17/Th22-related cytokines will be assayed to determine the mechanisms of the anti-inflammatory and immunomodulatory effects of the mixed CHF in AD patients. The nature of the microbiome dysfunction underlying this disease will be explored. Investigators will also apply a metabolomics approach to reveal the plasma metabolites in AD patients of different TCM patterns as well as to monitor changes of plasma metabolome in AD patients under mixed CHF treatment, aiming to develop metabolic biosignatures for efficacy of mixed CHF in AD patients exhibiting specific TCM pattern. PK study will be conducted to exam blood concentration of the prescription in healthy volunteers and AD patients with good or poor drug response. The results will provide evidence for the precision treatment based on different TCM pattens of AD patients. Completion of this integrated project will provide innovative information for future clinical applications.

DETAILED DESCRIPTION:
In this study, a randomized, double-blinded, placebo control trial is designed and total 120 AD patients will be enrolled. All participants will be divided into Chinese herbal formula (CHF) and placebo control groups, in 2:1 allocation ratio. CHF group will receive capsules of mixture CHF; while control group will receive placebo capsules with similar look, smell, and taste with same scheme. Total 12-week treatment course will be done.

Aim 1: The effects and immunomodulatory mechanisms of a mixed CHF in AD patients with different TCM patterns

1A: Measurement of AD severity by Scoring of AD (SCORAD) scale and assessment of health-related quality of life using the Dermatology Life Quality Index (DLQI) or Children's Dermatology Life Quality Index (CDLQI)

1B: Reduction rate of exposure to western medicine after a mixed CHF treatment

1C: The effects of CHF treatment on CRP, ESR, eosinophil count, IgE, CD4+/CD8+ and related cytokines / signaling pathway involved in AD regulation

1. D: Safety evaluation by measuring side effects, hemogram, electrolytes, kidney and liver function Aim 2: Effects of a mixed CHF on gut microbiota in AD patients
2. A: Fecal DNA purification and 16S rRNA gene sequencing before and after CHF treatment

2B: Bioinformatics analysis to explore microbial dysfunction underlying AD and changes of gut microbiome after CHF treatment 2C: Determination of short-chain fatty acid (SCFA) levels in fecal samples before and after CHF treatment Aim 3: Effects of a mixed CHF on plasma metabolomes of AD patients 3A: Plasma metabolomics analysis in AD patients with different TCM patterns 3B: Plasma metabolomics analysis in AD patients under a mixed CHF treatment 3C: Determination of the previously known immunomodulatory metabolites in AD patients under a mixed CHF treatment Aim 4: PK study between healthy volunteers, valid patients, and patients with poor response to the mixed CHF 4A: Preparation and quality control of target prescription 4B: PK study of the mixed CHF

ELIGIBILITY:
Inclusion Criteria:

1. All volunteers must sign an informed consent form.
2. Male and female patients aged 6 to 60 years.
3. Patients who are diagnosed with AD by expert clinicians at Taoyuan, Linkou or Taipei Chang Gung Memorial Hospital and Taipei Veterans General Hospital in Taiwan and met the criteria of Hanifin and Rajka diagnostic criteria will be considered for enrollment in this study.
4. SCORing Atopic Dermatitis (SCORAD) score ≧ 25

Exclusion Criteria:

1. Other skin diseases that are not AD, such as contact dermatitis, seborrheic dermatitis, or drug-induced dermatitis, which will be diagnosed by expert clinicians
2. Patients with other itching skin diseases at the same time, diagnosed by expert clinicians
3. Patients who have secondary bacterial infections or receiving oral or intravenous steroid treatment, antibiotics, leukotriene modifiers, phototherapy or other immunosuppressive therapies in the previous 1 month
4. Patients who cannot take the medicine regularly, or who can not cooperate in writing the questionnaires or taking blood tests
5. Allergy to Chinese medicine or use of other Chinese medicine treatments
6. Severe organ dysfunction, such as impaired renal and hepatic function at initial diagnosis (including chronic kidney disease stages III, IV, and V and AST, ALT ≥3 × the upper normal limit), liver cirrhosis, or heart failure
7. Uncontrolled psychiatric problems or other severe systemic diseases
8. Current pregnant or breast-feeding women, and all women of childbearing age must agree to take appropriate contraceptive precautions

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes of SCORing Atopic Dermatitis (SCORAD) score after treatment with a mixed CHF (composed of Xiao-Feng-San + Zhen-Ren-Huo-Ming-Yin + Dictamnus dasycarpus + Houttuynia cordata) | Assess at the beginning of the study and after 6 and 12 weeks' treatment, total 3 times
  Measurement of symptoms related to AD including the severity of eczema, pruritis, and insomnia. The score ranges from 0 to 103 and higher scores mean a worse outcome.
Changes of Dermatology Life Quality Index (DLQI) score (use Children's Dermatology Life Quality Index, CDLQI, for patients at the ages of 6 to 16 years) after treatment with a mixed CHF | Assess at the beginning of the study and after 6 and 12 weeks' treatment, total 3 times
  Measurement of quality of life.The score ranges from 0 to 30 and higher scores mean a worse outcome.
Changes of exposure to western medicine by recording the name and dosage of western medicine used for AD treatment | Assess at the beginning of the study, then weekly, up to 12 weeks
  To explore whether the use of western medicine could be reduced after treatment with a mixed CHF

SECONDARY OUTCOMES:
Changes of ESR level after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Evaluation of serologic markers related to AD
Changes of CRP level after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Evaluation of serologic markers related to AD
Changes of eosinophil count after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Evaluation of serologic markers related to AD
Changes of IgE level after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Evaluation of serologic markers related to AD
Changes of CD4/CD8 ratio after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Evaluation of serologic markers related to AD
Changes of IL-4, IL-5, IL-10, IL-12, IL-13, IL-17, IL-22, IL-23, and INF-γ level after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Evaluation of serologic markers related to AD
Changes of JAK1, JAK2, JAK3, tyrosine kinase-2 (TYK2), STAT1, STAT2, STAT3, STAT4, and STAT5 level after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Evaluation of JAK-STAT signaling pathway
Changes of gut microbiota | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  Differences of gut microbiota in AD patients with different TCM patterns before and after treatment and the effects of altered gut microbial colonization on the severity of AD
Differences in the AD-associated metabolites (phosphatidylcholine, acylcarnitine) between AD patients with different TCM patterns after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  To investigate whether plasma concentrations of these known metabolites are associated with the efficacy of a mixed CHF treatment in AD patients
Differences in the anti-inflammatory metabolites (itaconate and its derivative, 4-octyl itaconate) between AD patients with different TCM patterns after a mixed CHF treatment | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  To investigate whether plasma concentrations of these known metabolites are associated with the efficacy of a mixed CHF treatment in AD patients
Compare blood concentration of mixed CHF between AD patients with different TCM patterns after a mixed CHF treatment by PK study | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  The maximal measured plasma concentration (Cmax) will be taken
Concentration-time profile of mixed CHF between AD patients with different TCM patterns after a mixed CHF treatment by PK study | Assess at the beginning of the study and after 12 weeks' treatment, total 2 times
  The time at which the maximal plasma concentration observed (Tmax) will be taken from the observed plasma concentration-time profile